CLINICAL TRIAL: NCT05522335
Title: A Phase III Randomized Open Label Multi-center Study to Compare Immunogenicity and Safety of BBV154 With COVAXIN®, and to Assess Lot to Lot Consistency of BBV154 in Healthy Volunteers
Brief Title: Phase III Study of BBV154 Intranasal Vaccine in Healthy Volunteers
Acronym: Nasal154PH3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BBIL/BBV154-III/2022; BBIL/BBV154-III/2022 (Other: Bharat Biotech International limited)
Record Dates: First submitted 2022-08-13; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — BBV152 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BBV154 Lot-1 (Active Comparator): Safety Group : In this group, 1000 participants will be recruited, receive BBV154 vaccine (0.5 mL each dose) on day 0 and day 28 via intranasal route and assess for the safety.
  Interventions: Biological: BBV154(Intranasal) & covaxin
- BBV154 Lot-2 (Active Comparator): Safety Group : In this group, 1000 participants will be recruited, receive BBV154 vaccine (0.5 mL each dose) on day 0 and day 28 via intranasal route and assess for the safety.
  Interventions: Biological: BBV154(Intranasal) & covaxin
- BBV154 Lot-3 (Active Comparator): Safety Group : In this group, 1000 participants will be recruited, receive BBV154 vaccine (0.5 mL each dose) on day 0 and day 28 via intranasal route and assess for the safety.
  Interventions: Biological: BBV154(Intranasal) & covaxin
- COVAXIN® (Active Comparator): Immunogenicity Group :In this group, 160 participants will be recruited, receive Covaxin vaccine (0.5 mL each dose) on day 0 and day 28 via intramuscular route and assess for the Immunogenicity.
  Interventions: Biological: BBV154(Intranasal) & covaxin

INTERVENTIONS:
Biological: BBV154(Intranasal) & covaxin — Intervention Covaxin

SUMMARY:
Group 1 (BBV154): In this group, 3000 participants will be recruited, randomized in 1:1:1 ratio receive 3 consecutive lots (Lot 1: 1000, Lot 2: 1000, Lot 3: 1000) of the BBV154 vaccine (0.5 mL each dose) on day 0 and day 28 via intranasal route. Group 2 (COVAXIN®): In this group, 160 participants will be recruited and administered with COVAXIN® vaccine on day 0 and on day 28 via intramuscular route.

A total sample size of 3160 healthy volunteer's age's ≥18 years will be recruited in this study. BBV154-Subjects- Part 1 ( Immunogenicity Group)- First 640 Subjects BBV154-Subjects- Part 2 ( Safety Group)- (Remaining 2520 subjects) Visit 1: Baseline (Day 0) Visit 2 (Day 28+2) Visit 3 (Day 42 ± 7 days) Visit 4 (Day 90 ± 7 days) and Visit 5 (Day 180± 7 days)

DETAILED DESCRIPTION:
Sample Collection:

1. Pregnancy test will be conducted by using rapid test kit.
2. Immunogenicity analysis: A total of 5 ml of blood is collected on Day 0, Day 28+2, Day 42±7, Day 90±7 and Day 180±7 (Subset of 640, 160 from each lot and control group). Sera will collect from the blood sample and stored as 3 aliquots at -20°C.
3. A saliva sample (5 mL) and an additional blood sample (10mL) will be collected on Day 0, Day 28+2, Day 42±7, Day 90±7 and Day 180±7 (Subset of 80, 60 from Group 1(20 from each lot) and 20 from Group 2).
4. Saliva will be collected by Passive droll method using Falcon tube.

Sample Size:

A total sample size of 3160 healthy volunteer's age's ≥18 years will be recruited in this study.

Randomization:

A total of 3000 participants will be randomized in to BBV154 two-dose study arm and 160 participants in the COVAXIN® two-dose arm. The first 640 participants are randomized with block size 4, in 1:1:1:1 ratio [(3 (BBV154): 1 (COVAXIN®)].

Remaining 2520 participants in the study are randomized with the block size 6 in 1:1:1 ratio (BBV154).

STUDY RATIONALE:

Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection is accelerating globally, leading to an increase in morbidity and mortality. The high-risk group includes the health care workers (HCW) (physicians and paramedical staff), working amid SARS-CoV-2 infected patients, all other people including household contacts of COVID-19 confirmed patients, people currently residing or working in COVID-19 hot-spots/outbreak areas where there is a high risk of transmission of SARS-CoV-2 infection and especially the elderly people (age >60 Years). Though SARS-CoV-2 infection may cause mild symptoms in many, nearly 14% develop severe disease that requires hospitalization and oxygen support, and 5% require admission to an intensive care unit (ICU). In severe cases, COVID-19 can be complicated by acute respiratory distress syndrome, sepsis, septic shock, and multi organ failure (2,3).

Though the antiviral drugs such as Remdesivir has been approved for COVID-19 treatment by USFDA, but it fails to prevent COVID-19 deaths (3). Hence, there is a necessity to develop a vaccine to prevent SARS-CoV-2 infection. Various types of COVID-19 vaccines, such as DNA, RNA based formulations, recombinant subunit vaccines containing the viral protein (Spike) epitopes, vector-based mutations (eg: Adenovirus and traditional inactivated vaccines are under development(6-9). A chimpanzee adenoviral vaccine (Adenoviral vectored-SARS-CoV-2-S), encoding prefusion stabilized spike protein of SARS-CoV-2 virus was developed by Washington University School of Medicine, and evaluated the protective activity of the vaccine in challenge studies with SARS-CoV-2 virus and mice expressing human angiotensin-converting enzyme 2 (ACE2) receptor(10). Challenge study results were revealed that intramuscular dosing of Adenoviral vectored-SARS-CoV-2-S vaccine induces systemic humoral and cell mediated immunity and protects against lung infection whereas intranasal dosing of the same vaccine induces both systemic and mucosal immunoglobulins (IgG and IgA) ad protects from lower and upper respiratory tract infections (10). Bharat Biotech has collaborated with Washington University to manufacture the vaccine and conduct clinical trials.

BBV154 intranasal vaccine was evaluated for its safety and immunogenicity in a Phase 1 clinical study in 175 healthy participants and found to be safe and immunogenic with two dose regimen administered with 4 weeks interval. In a Phase 2/3 clinical study, BBV154 vaccine with two dose regimen is further evaluating in 152 participants for its safety and immunogenicity. Bharat Biotech has designed this pivotal Phase 3 study to immunogenicity, safety and lot- to-lot consistency of the BBV154 vaccine compared to COVAXIN® vaccine.

STUDY DESIGN:

The Phase-III study is designed to evaluate the immunogenicity, safety and lot-to-lot consistency of two groups of healthy volunteers who receive either BBV154 vaccine via intranasal route or COVAXIN® vaccine via intramuscular route. A total of 3160 participants will be enrolled and assess for the safety, immunogenicity and lot consistency.

Group 1 (BBV154): In this group, 3000 participants will be recruited, randomized in 1:1:1 ratio receive 3 consecutive lots (Lot 1: 1000, Lot 2: 1000, Lot 3: 1000) of the BBV154 vaccine (0.5 mL each dose) on day 0 and day 28 via intranasal route.

Group 2 (COVAXIN®): In this group, 160 participants will be recruited and administered with COVAXIN® vaccine on day 0 and on day 28 via intramuscular route.

STUDY PROCEDURES

Visit 1: Baseline (Day 0):

1. The participant will be screened for eligibility based on medical history, vitals, and physical examination and urine pregnancy test for female participants.
2. If the participant is eligible (in good general health or stable pre-existing disease as per the discretion of the Principal investigator), a blood sample will be withdrawn prior to vaccination (Subset).
3. Blood sample (5 mL) will be collected from subset (n=640, 160 from each lot of Group 1 & Group 2) of participants.
4. Saliva sample (5 mL) will be collected from subset (n=80, 60 from Group 1 (20 from each lot) and 20 from Group 2) of participants.
5. An additional 10 mL of blood sample will be collected from subset (n=80, 60 from Group 1 (20 from each lot) and 20 from Group 2) of participants.
6. An intranasal vaccine or COVAXIN® will be administered. Following vaccination, participants will remain at the study site for at least 30 minutes of observation to record any immediate adverse event.
7. Diary card will be distributed to the participants.
8. Telephonic follow-up (7-days post-vaccination) for adverse event recording.

   Visit 2 (Day 28+2):
9. Study participants will return to the OPD for vitals and physical examination (general and systemic examination and urine pregnancy test for female participants), and specific symptoms for COVID-19.
10. Blood sample (5 mL) will be collected from subset (n=640, 160 from each lot of Group 1 & Group 2) of participants.
11. Saliva sample (5 mL) will be collected from subset (n=80, 60 from Group 1(20 from each lot) and 20 from Group 2) of participants.
12. An additional 10 mL of blood sample will be collected from subset (n=80, 60 from Group 1(20 from each lot) and 20 from Group 2) of participants.
13. An intranasal vaccine or COVAXIN® will be administered. Following vaccination, participants will remain at the study site for at least 30 minutes of observation to record any adverse event.
14. Diary card will be collected and a new diary card distributed to the participants.
15. Telephonic follow-up (7-days post-vaccination) for adverse event recording.

Visit 3 (Day 42 ± 7 days):

1. Study participants will return to the OPD for physical examination (general and systemic examination and urine pregnancy test for female participants), and specific symptoms for COVID-19.
2. Blood sample (5 mL) will be collected from subset (n=640, 160 from each lot of Group 1 & Group 2) of participants.
3. Saliva sample (5 mL) will be collected from subset (n=80, 60 from Group 1(20 from each lot) and 20 from Group 2) of participants.
4. An additional 10 mL of blood sample will be collected from subset (n=80, 60 from Group 1(20 from each lot) and 20 from Group 2) of participants.
5. Diary card will be collected from the participants.

Visit 4 (Day 90 ± 7 days):

1. Study participants (Subset) will return to the OPD for physical examination (general and systemic examination), and specific symptoms for COVID-19.
2. Urine pregnancy test for female participants (Immunogenicity subset)
3. Blood sample (5 mL) will be collected from subset (n=640, 160 from each lot of Group 1 & Group 2) of participants.
4. Saliva sample (5 mL) will be collected from subset (n=80, 60 from Group 1(20 from each lot) and 20 from Group 2) of participants.

4. An additional 10 mL of blood sample will be collected from subset (n=80, 60 from Group 1(20 from each lot) and 20 from Group 2) of participants.

5. Safety data will be collected from all the participants through telephonically other than immunogenicity subset (Day 90 ± 7 days).

Visit 5 (Day 180± 7 days):

1. Study participants (Subset) will return to the OPD for physical examination (general and systemic examination), and specific symptoms for COVID-19.
2. Urine pregnancy test for female participants (Immunogenicity subset)
3. Blood sample (5 mL) will be collected from subset (n=640, 160 from each lot of Group 1 & Group 2) of participants.
4. Saliva sample (5 mL) will be collected from subset (n=80, 60 from Group 1(20 from each lot) and 20 from Group 2) of participants.
5. An additional 10 mL of blood sample will be collected from subset (n=80, 60 from Group 1 (20 from each lot) and 20 from Group 2) of participants.
6. Safety data will be collected from all the participants through telephonically other than immunogenicity subset (Day 180 ± 7 days).

Safety Monitoring:

Subjects will be observed for 30 minutes after vaccination for immediate adverse events. Active surveillance will be conducted for all participants for seven days after each dose of vaccine to ascertain information on solicited adverse events ("Reactogenicity"). Safety data will be collected from all the participants through telephonically on Day 90± 7 and 180± 7.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent.
2. Participants of either gender of age ≥18 years.
3. Good general health as determined by the discretion of investigator (vital signs (heart rate ≥60 to≤100 bpm; blood pressure systolic ≥90 mm Hg and <140 mm Hg; diastolic ≥ 60 mm Hg and <90 mm Hg; oral temperature <100.4ºF), medical history, and physical examination).
4. Expressed interest and availability to fulfill the study requirements.
5. For a female participant of child-bearing potential, planning to avoid becoming pregnant (use of an effective method of contraception or abstinence) from the time of study enrolment until at least four weeks after the last vaccination
6. Male subjects of reproductive potential: Use of condoms to ensure effective contraception with the female partner from first vaccination until 3 months after last vaccination
7. Participants must refrain from blood/plasma or any other bodily fluid donation from the time of first vaccination until 3 months after last vaccination
8. Agrees not to participate in another clinical trial at any time during the study period.
9. Agrees to remain in the study area for the entire duration of the study.
10. Willing to allow storage and future use of biological samples (serum) for future research.

    -

Exclusion Criteria:

1. History of any other COVID-19 investigational/or licensed vaccination.
2. For women of child bearing potential, a positive serum pregnancy test (during screening within 45 days of enrolment) or positive urine pregnancy test (within 24 hours of administering each dose of vaccine).
3. Temperature >38.0°C (100.4°F) or symptoms of an acute self limiting illness such as an upper respiratory infection or gastroenteritis within three days prior to each dose of vaccine.
4. Medical problems because of alcohol or illicit drug use during the past 12 months.
5. Receipt of an experimental agent (vaccine, drug, device, etc.) within 60 days before enrolment or expects to receive an investigational agent during the study period.
6. Receipt of any licensed vaccine (other than Covid-19 vaccine) within four weeks before enrolment in this study.
7. Known sensitivity to any ingredient of the study vaccines, or a more severe allergic reaction and history of allergies in the past.
8. Receipt of immunoglobulin or other blood products within the three months prior to vaccination in this study.
9. Immunosuppressant as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
10. Long-term use (> 2 weeks) of oral or parenteral steroids (glucocorticoids) or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding six months (Topical steroids are allowed).
11. Any history of anaphylaxis in relation to vaccination.
12. History of any cancer.
13. History of severe psychiatric conditions likely to affect participation in the study.
14. A bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder, or prior history of significant bleeding or bruising following IM injections or venepuncture).
15. Any other serious chronic illness requiring immediate hospital specialist supervision.
16. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3160 (Actual)
Dates: Start 2022-04-16 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titres (GMTs | baseline
  Serum neutralising antibody titer (NAb"s) by neutralizing antibody assays.
Geometric mean titres (GMTs | Day 28+2
  Serum neutralising antibody titer (NAb"s) by neutralizing antibody assays.
Geometric mean titres (GMTs) | Day 42±7
  Serum neutralising antibody titer (NAb"s) by neutralizing antibody assays
Geometric mean titres (GMTs) | Day 90±7
  Serum neutralising antibody titer (NAb"s) by neutralizing antibody assays
Geometric mean titres (GMTs) | Day 180±7.
  Serum neutralising antibody titer (NAb"s) by neutralizing antibody assays
solicited adverse events | 7days
  The occurrence of solicited adverse events within seven days of vaccination
unsolicited adverse events | day 180
  The occurrence of any unsolicited adverse events up to day 180 from 1st dose vaccination.

SECONDARY OUTCOMES:
Geometric mean titers (GMTs) | baseline
  salivary IgA (n=80), Serum IgA and IgG binding antibody titer by ELISA assays
Geometric mean titers (GMTs) | Day 28+2
  salivary IgA (n=80), Serum IgA and IgG binding antibody titer by ELISA assays
Geometric mean titers (GMTs) | Day 42±7
  salivary IgA (n=80), Serum IgA and IgG binding antibody titer by ELISA assays
Geometric mean titers (GMTs) | Day 90±7
  salivary IgA (n=80), Serum IgA and IgG binding antibody titer by ELISA assays
Geometric mean titers (GMTs) | Day 180±7
  salivary IgA (n=80), Serum IgA and IgG binding antibody titer by ELISA assays
Geometric mean titres | baseline
  Serum neutralising antibody titer (NAb"s) by neutralizing antibody assays.
Geometric mean titres | Day 28+2
  Serum neutralising antibody titer (NAb"s) by neutralizing antibody assays.
Geometric mean titres | Day 42±7
  Serum neutralising antibody titer (NAb"s) by neutralizing antibody assays.
adverse event | 180 Days
  The occurrence of adverse event of special interest (AESI).
vaccine induced thrombosis and thrombocytopenia | 180 Days
  The occurrence of the vaccine induced thrombosis and thrombocytopenia in participants reporting the respective symptoms and signs.

CONTACTS AND LOCATIONS:
Locations (14):
- India (14):
  - VIMS (Visakha Institute of Medical Sciences), Vizag, Andhrapradesh
  - AIIMS (All India Institute of Medical Sciences), Patna, Bihar
  - Redkar Hospital and Research center, Dargalim, Goa
  - Aatman Hospital, Ahmedabad, Ahmedabad, Gujarat
  - PGIMS (Pt. BD Sharma Postgraduate Institute of Medical Sciences), Rohtak, Haryana
  - Jeevan Rekha Hospital, Belgaum, Belagavi, Karnataka
  - Rajarajeshwari Medical College and Hospital, Kambīpura, Karnataka
  - Oyster and Pearl Hospitals (Phadnis Clinic Pvt Ltd), Pune, Maharashtra
  - Acharya Vinobha Bhave Rural Hospital, Wardha, Maharashtra
  - Maharaja Agrasen super specality Hospital, Jaipur, Jaipur, Rajasthan
  - Malla Reddy Narayana Multi Speciality Hospital, Hyderabad, Telangana
  - NIMS (Nizam's Institute of Medical Sciences, Hyderabad, Telangana
  - Rana Hospital, Gorakhpur, Uttar Pradesh
  - Prakhar Hospital, Kanpur, Uttar Pradesh

REFERENCES:
- [Derived] Singh C, Verma S, Reddy P, Diamond MS, Curiel DT, Patel C, Jain MK, Redkar SV, Bhate AS, Gundappa V, Konatham R, Toppo L, Joshi AC, Kushwaha JS, Singh AP, Bawankule S, Ella R, Prasad S, Ganneru B, Chiteti SR, Kataram S, Vadrevu KM. Phase III Pivotal comparative clinical trial of intranasal (iNCOVACC) and intramuscular COVID 19 vaccine (Covaxin(R)). NPJ Vaccines. 2023 Aug 18;8(1):125. doi: 10.1038/s41541-023-00717-8. PMID 37596281
- [Derived] Nakahashi-Ouchida R, Fujihashi K, Kurashima Y, Yuki Y, Kiyono H. Nasal vaccines: solutions for respiratory infectious diseases. Trends Mol Med. 2023 Feb;29(2):124-140. doi: 10.1016/j.molmed.2022.10.009. Epub 2022 Nov 23. PMID 36435633